CLINICAL TRIAL: NCT05034900
Title: Does Addition of Oscillatory Positive Expiratory Pressure (OPEP) Device to a Chest Physiotherapy Program Provide Further Health Benefits in Children With Bronchiectasis?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Melih Zeren, Assist. Prof. Dr., Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: bakircaymzeren05
Record Dates: First submitted 2021-09-01; First posted 2021-09-05 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Bronchiectasis
Keywords: bronchiectasis; children; oscillatory positive expiratory pressure device; chest physiotherapy; pulmonary function; exercise capacity
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chest Physiotherapy Group (Active Comparator): Patients in this group will perform comprehensive chest physiotherapy program two times a day, 7 days a week for 8 weeks at their homes.
  Interventions: Other: Chest physiotherapy
- OPEP device + Chest Physiotherapy Group (Experimental): In addition to the same physiotherapy program applied to the controls, patients in this group will also use OPEP device two times a day, 7 days a week for 8 weeks at their homes.
  Interventions: Other: Chest physiotherapy; Device: Oscillatory Positive Expiratory Pressure (OPEP) device

INTERVENTIONS:
Other: Chest physiotherapy — Programme will include diaphragmatic breathing exercise, thoracic expansion exercises, postural drainage and coughing techniques.
Device: Oscillatory Positive Expiratory Pressure (OPEP) device — Shaker® device will be used.
  Arms: OPEP device + Chest Physiotherapy Group

SUMMARY:
Oscillatory positive expiratory pressure (OPEP) devices such as Flutter®, Aerobika® or Shaker ® are commonly prescribed in the clinical practice for airway clearance in children with chronic lung diseases including bronchiectasis, cystic fibrosis, and primary ciliary dyskinesia. Health insurance companies may cover these devices in some countries; but this is not a common practice around the world. Therefore, many families have to purchase these devices themselves. Unfortunately, these devices are rather expensive especially in the developing countries and consequently, families become financially burdened. Aim of this study is to investigate whether the addition of OPEP devices to a comprehensive chest physiotherapy program provide additional benefits on pulmonary function and exercise capacity in children with bronchiectasis. Results of this study may help better interpreting the cost-effectiveness of these devices.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bronchiectasis

Exclusion Criteria:

* Hospitalization history during past month
* Diagnosis of any other chronic childhood diseases such as cerebral palsy or neuromuscular diseases which may impede exercise tolerance

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline Forced Vital Capacity (FVC) at 8 weeks | 8 weeks
  Forced Vital Capacity (FVC) will be measured using Spiropalm 6MWT device
Change from baseline Forced Expiratory Volume in 1 second (FEV1) at 8 weeks | 8 weeks
  Forced Expiratory Volume in 1 second (FEV1) will be measured using Spiropalm 6MWT device
Change from baseline Peak Expiratory Flow (PEF) at 8 weeks | 8 weeks
  Peak Expiratory Flow (PEF) will be measured using Spiropalm 6MWT device
Change from baseline maximum minute ventilation at 8 weeks | 8 weeks
  Maximum minute ventilation will be measured using Spiropalm 6MWT device during six-minute walk test
Change from baseline breathing reserve at 8 weeks | 8 weeks
  Breathing reserve will be measured using Spiropalm 6MWT device during six-minute walk test
Change from baseline six-minute walk distance at 8 weeks | 8 weeks
  Distance walked in six minutes will be recorded in six-minute walk test.
Change from baseline M. Quadriceps strength at 8 weeks | 8 weeks
  M. Quadriceps strength will be measured using hand-held dynamometer
Change from baseline Leicester Cough Questionnaire score at 8 weeks | 8 weeks
  Questionnaire consists of 19 items covering physical, psychological and social domains of chronic cough with a 7 point likert response scale (range from 1 to 7). Higher score indicates better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Faculty of Medicine, Department of Pediatrics, Division of Pediatric Pulmonology, Izmir, Turkey (Türkiye)